CLINICAL TRIAL: NCT02966028
Title: A Double-blind, Randomised, Placebo-controlled Study to Assess the Effect of SNF472 on Progression of Cardiovascular Calcification on Top of Standard of Care in End-stage-renal-disease (ESRD) Patients on Hemodialysis (HD)
Brief Title: Effect of SNF472 on Progression of Cardiovascular Calcification in End-Stage-Renal-Disease (ESRD) Patients on Hemodialysis (HD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanifit Therapeutics S. A. (Other)
Collaborators: Clinipace Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNFCT2015-05
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Results first posted 2021-03-16 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Diseases; Cardiovascular Abnormalities; Calcifications, Vascular; Endstage Renal Disease; ESRD; Coronary Artery Calcification
Keywords: CAC; calcium; ESRD; calcification; cardiovascular; heart; kidney; hemodialysis; Agatston
MeSH Terms: conditions — Cardiovascular Diseases; Cardiovascular Abnormalities; Vascular Calcification; Kidney Failure, Chronic; Calcinosis | interventions — SNF472

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SNF472 300 mg (Experimental): Dose 1 arm (300 mg): 1 vial of physiological saline and 1 vial of active (10 mL SNF472 at 30 mg/mL)
  Interventions: Drug: SNF472
- SNF 472 600 mg (Experimental): Dose 2 arm (600 mg): 2 vials of active (10 mL SNF472 at 30 mg/mL)
  Interventions: Drug: SNF472
- Matching Placebo (Placebo Comparator): Placebo arm: 2 vials of physiological saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SNF472 — Administered 3 times weekly by intravenous infusion through the dialysis machine in conjunction with the patient's dialysis sessions.
  Arms: SNF 472 600 mg; SNF472 300 mg
Drug: Placebo — Administered 3 times weekly by intravenous infusion through the dialysis machine in conjunction with the patient's dialysis sessions.
  Arms: Matching Placebo

SUMMARY:
The primary objective is to assess the effect of 2 dose levels of SNF472 (300 mg and 600 mg) compared to placebo on the progression of coronary artery calcium volume score over a 12-month (52 weeks) period in ESRD patients on HD

DETAILED DESCRIPTION:
Reducing the progression of cardiovascular calcification (CVC) in HD patients may improve the severe burden of CV disease related to the underlying ESRD. As no therapy is currently indicated to target CVC, there is a need to investigate the ability of SNF472 to reduce CVC progression and, ultimately, to improve CV outcomes in HD patients. This phase 2b double-blind, randomised, placebo-controlled study is designed to assess the effect of SNF472 on the progression of CVC as measured by calcium volume and CAC/Agatston scores in ESRD patients receiving HD. The study hypothesis is that administration of SNF472 over 52 weeks can slow the progression of CVC in this patient population compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients, 18 to 80 years (inclusive) of age at randomisation
* CAC score of 100 to 3500 AU (Agatston Units) inclusive within a 3-week period prior to randomisation as measured by a multi-detector CT scanner
* Patients who are EITHER ≥ 55 years OR have a history of diabetes mellitus at randomisation
* Patients on HD for ≥ 6 months prior to randomisation
* Willing and able to understand and sign the informed consent

Exclusion Criteria:

* Scheduled date for kidney transplant from a known living donor
* Weight above 300 lbs (136 kg)
* Hospitalisation in the previous 3 months prior to randomisation for unstable angina, MI, stroke, transient ischaemic attack, amputation or peripheral or coronary bypass surgery
* History of unstable heart failure in the previous 3 months, defined as an unplanned presentation to a hospital or dialysis treatment facility with signs/symptoms of acute pulmonary edema and requiring ultrafiltration therapy
* History of cancer that has been in remission for < 5 years prior to randomisation. A history of basal cell carcinoma or Stage 1 squamous cell carcinoma of the skin is allowed
* Pregnant or trying to become pregnant, currently breast-feeding, or of child-bearing potential (including peri-menopausal women who have had a menstrual period within one year) and not willing to practice birth control using a double barrier method (criteria apply to women only) at least 30 days post last dose of study medication
* Hypocalcaemia defined as a serum calcium below 8.0 mg/dL (or 2.0 mmol/L) for the serum calcium most proximal to screening per patient's medical records
* Extreme elevation in serum phosphorous, defined as a serum phosphorous above 10 mg/dL (or 3.23 mmol/L) within the last 2 months proximal to screening per patient's medical records
* Uncontrolled hypertension defined as any 2 or more consecutive post-dialysis diastolic blood pressure (DBP) > 100 mmHg within the last 2 months proximal to screening expected survival < 2 years in the Investigator's medical opinion
* Known active drug or alcohol abuse within 1 year of randomisation
* Use of other investigational drugs within 30 days of randomisation
* Non-compliance with dialysis treatment which, in the opinion of the Investigator, evidenced by either repeated missed dialysis treatments or significant non-compliance with the patient's medication regimen
* Inability to comply with all required study procedures and schedule, inability to speak and read in the protocol-derived language of that patient's clinical site, or unwillingness or inability to give written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2016-11; Primary Completion 2019-08 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Gold, MD, Study Director — Sanifit Chief Medical Officer
Locations (67):
- United States (45):
  - Bakersfield, California
  - Chula Vista, California
  - Escondido, California
  - Granada Hills, California
  - La Palma, California
  - Long Beach, California
  - Los Angeles, California
  - Lynwood, California
  - Northridge, California
  - Riverside, California
  - San Diego, California
  - San Dimas, California
  - Simi Valley, California
  - Tarzana, California
  - Whittier, California
  - Arvada, Colorado
  - Westminster, Colorado
  - Middlebury, Connecticut
  - Orange, Connecticut
  - Hollywood, Florida
  - Lauderdale Lakes, Florida
  - Miami, Florida
  - Miami Gardens, Florida
  - Ocala, Florida
  - Tampa, Florida
  - Evanston, Illinois
  - Shreveport, Louisiana
  - Pontiac, Michigan
  - Roseville, Michigan
  - Brookhaven, Mississippi
  - Las Vegas, Nevada
  - Reno, Nevada
  - North Brunswick, New Jersey
  - College Point, New York
  - The Bronx, New York
  - Asheville, North Carolina
  - Cincinnati, Ohio
  - Bethlehem, Pennsylvania
  - Knoxville, Tennessee
  - Arlington, Texas
  - Houston, Texas
  - Richardson, Texas
  - San Antonio, Texas
  - Chesapeake, Virginia
  - Wauwatosa, Wisconsin
- Spain (16):
  - Palma, Balearic Islands
  - Palma de Mallorca, Balearic Islands
  - Barcelona, Catalonia
  - Galdakao, Vizcaya
  - Barcelona
  - Córdoba
  - Lleida
  - Lugo
  - Madrid
  - Navarro
  - Oviedo
  - Palma
  - Santander
  - Seville
  - Valencia
  - Zaragoza
- United Kingdom (6):
  - Bradford
  - Manchester
  - Salford
  - Shrewsbury
  - Swansea
  - Westcliff-on-Sea

REFERENCES:
- [Derived] Perello J, Alberti J, Torres JV, Ferrer MD, Perez MM, Bassissi F, Gold A, Raggi P, Chertow GM, Salcedo C. Hexasodium fytate exposure-response correlations in a randomized, placebo-controlled study of patients on dialysis with cardiovascular calcification. Front Pharmacol. 2024 Feb 7;15:1325186. doi: 10.3389/fphar.2024.1325186. eCollection 2024. PMID 38384289
- [Derived] Bushinsky DA, Raggi P, Bover J, Ketteler M, Bellasi A, Rodriguez M, Sinha S, Garg R, Perello J, Gold A, Chertow GM; CaLIPSO Investigators*; CaLIPSO Study Group and Clinipace GmbH, Intrinsic Imaging, LLC. Effects of Myo-inositol Hexaphosphate (SNF472) on Bone Mineral Density in Patients Receiving Hemodialysis: An Analysis of the Randomized, Placebo-Controlled CaLIPSO Study. Clin J Am Soc Nephrol. 2021 May 8;16(5):736-745. doi: 10.2215/CJN.16931020. Epub 2021 Apr 7. PMID 33835939
- [Derived] Raggi P, Bellasi A, Bushinsky D, Bover J, Rodriguez M, Ketteler M, Sinha S, Salcedo C, Gillotti K, Padgett C, Garg R, Gold A, Perello J, Chertow GM. Slowing Progression of Cardiovascular Calcification With SNF472 in Patients on Hemodialysis: Results of a Randomized Phase 2b Study. Circulation. 2020 Mar 3;141(9):728-739. doi: 10.1161/CIRCULATIONAHA.119.044195. Epub 2019 Nov 11. PMID 31707860

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SNF472 300 mg | SNF 472 600 mg | Matching Placebo
Started | 92 | 91 | 91
Completed | 68 | 57 | 60
Not Completed | 24 | 34 | 31
Not completed — Adverse Event | 7 | 13 | 10
Not completed — Physician Decision | 1 | 0 | 2
Not completed — Withdrawal by Subject | 7 | 5 | 5
Not completed — Kidney transplant Changed dialysis units | 9 | 16 | 14

BASELINE CHARACTERISTICS:
Population: One subject randomized to placebo discontinued from the trial prior to the initiation of the study drug. The number of subjects treated and analyzed was 273 and the number of subjects randomized was 274.
Groups:
- Total: Total of all reporting groups
Arm/Group | SNF472 300 mg | SNF 472 600 mg | Matching Placebo | Total
Number analyzed (Participants) | 92 | 91 | 90 | 273
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 54 | 51 | 40 | 145
  >=65 years | 38 | 40 | 50 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9.5) | 64 (8.9) | 64. (8.2) | 63.5 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 36 | 33 | 107
  Male | 54 | 55 | 57 | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 36 | 32 | 99
  Not Hispanic or Latino | 60 | 51 | 56 | 167
  Unknown or Not Reported | 1 | 4 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 2 | 4 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 27 | 15 | 19 | 61
  White | 59 | 67 | 62 | 188
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 4 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 58 | 53 | 54 | 165
  United Kingdom | 6 | 3 | 5 | 14
  Spain | 28 | 35 | 31 | 94
CAC Agatston Score [Mean (Standard Deviation); unit: units on a scale] — Agatston score is a semi-automated tool to calculate a score the reflects the extent of coronary artery calcification as detected by an unenhanced CT scan. Scores range from 0 to >1000 Agatston units where higher scores indicate an increased amount of calcification and an increased risk for a major adverse cardiac event.
  units on a scale | 917 (697) | 963 (702) | 965 (762) | 948 (744)

OUTCOME MEASURES:

1. Primary Outcome: Change in Log CAC Volume Score From Baseline to Week 52 for the Combined Dose Groups vs Placebo
Description: Coronary Artery Calcification (CAC) Volume Score is a calculation to quantify the calcification of coronary artery calcium without factoring in the calcium density as measured by the CAC Agatston Score. The CAC Score was log-transformed and the primary outcome measure was the change in Log CAC Volume Score from Baseline to Week 52 for the combined dose groups vs placebo. The primary analysis used an ANCOVA model with the change in log volume score (log 52-week volume score - log baseline volume score) as the dependent variable and with a fixed effect term for the combined randomized treatment groups and log CAC volume score at baseline as a covariate. The least squares means for the treatment groups was estimated and back transformed.
  A smaller change from baseline to follow up is a better outcome.
Time Frame: Baseline (Week 1, Day 1) and Week 52
Population: Modified intent-to-treat (mITT) population, last observation carried forward (LOCF)
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Groups:
- SNF472 300 mg & 600 mg Combined: Dose (300 mg or 600 mg): 1 vial of physiological saline and 1 vial of active (10 mL SNF472 at 30 mg/mL) or 2 vials of active (10 mL SNF472 at 30 mg/mL)
  SNF472: Administered 3 times weekly by intravenous infusion through the dialysis machine in conjunction with the patient's dialysis sessions.
Arm/Group | SNF472 300 mg & 600 mg Combined | Matching Placebo
Number analyzed (Participants) | 142 | 77
ratio | 1.11 [1.067 to 1.153] | 1.20 [1.138 to 1.262]

2. Secondary Outcome: Change in Log CAC Volume Score From Baseline to Week 52 for Each Dose Group (300 mg and 600 mg) vs Placebo
Description: Coronary Artery Calcification (CAC) Volume Score is a calculation to quantify the calcification of coronary artery calcium without factoring in the calcium density as measured by the CAC Agatston Score. The CAC Score was log-transformed and the primary outcome measure was the change in Log CAC Volume Score from Baseline to Week 52 for the combined dose groups vs placebo. This secondary outcome measure was the change in Log CAC Volume Score from Baseline to Week 52 for each dose group vs placebo. The analysis used an ANCOVA model with the change in log volume score (log 52-week volume score - log baseline volume score) as the dependent variable and with a fixed effect term for each randomized treatment groups and log CAC volume score at baseline as a covariate. The least squares means for each of the treatment groups was estimated and back transformed.
  A smaller change from baseline to follow up is a better outcome.
Time Frame: Baseline (Week 1, Day 1) and Week 52
Population: Modified intent-to-treat (mITT) population, last observation carried forward (LOCF)
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | SNF472 300 mg | SNF 472 600 mg | Matching Placebo
Number analyzed (Participants) | 77 | 65 | 77
ratio | 1.12 [1.060 to 1.175] | 1.10 [1.042 to 1.165] | 1.20 [1.138 to 1.262]

3. Secondary Outcome: Change in Log CAC Agatston Score Between Baseline and Week 52 for Each Dose Group (300 mg and 600 mg) vs Placebo and for the Combined Dose Groups vs the Placebo Group
Description: Coronary Artery Calcification (CAC) Agatston Score is a semi-automated tool to calculate a score the reflects the extent of coronary artery calcification as detected by an unenhanced CT scan. Scores range from 0 to >1000 Agatston units where higher scores indicate an increased amount of calcification and an increased risk for a major adverse cardiac event. This secondary outcome measure was the change in Log CAC Agatston Score from Baseline to Week 52 for each dose group and the treated arms combined vs placebo. The analysis used an ANCOVA model with the change in log score (log 52-week score - log baseline score) as the dependent variable and with a fixed effect term for each randomized treatment groups and log CAC score at baseline as a covariate. The least squares means for each of the treatment groups separately and combined was estimated and back transformed.
Time Frame: Baseline (Week 1, Day 1) and Week 52
Population: Modified intent-to-treat (mITT) population, last observation carried forward (LOCF)
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Groups:
- SNF 472 Combined Dose Groups: Doses 300 and 600 mg. 1 vial of physiological saline and 1 vial of active or 2 vials of active(10 mL SNF472 at 30 mg/mL)
  SNF472: Administered 3 times weekly by intravenous infusion through the dialysis machine in conjunction with the patient's dialysis sessions.
Arm/Group | SNF472 300 mg | SNF 472 600 mg | SNF 472 Combined Dose Groups | Matching Placebo
Number analyzed (Participants) | 77 | 65 | 142 | 77
ratio | 1.10 [1.027 to 1.170] | 1.13 [1.055 to 1.215] | 1.11 [1.060 to 1.170] | 1.20 [1.122 to 1.278]

4. Secondary Outcome: Number of Subjects With <15% Progression in CAC Agatston Score From Baseline to Week 52 for Each Dose Group and the Combined Dose Groups vs Placebo
Description: Agatston score is a semi-automated tool to calculate a score that reflects the extent of coronary artery calcification as detected by an unenhanced CT scan. Scores range from 0 to >1000 Agatston units where higher scores indicate an increased amount of calcification and an increased risk for a major adverse cardiac event. Change in Agatston Score values from baseline to Week 52 were calculated as a percentage of change (progression or worsening of calcification). The number of subjects with <15% progression were counted.
Time Frame: Baseline (Week 1, Day 1) and Week 52
Population: Modified intent-to-treat (mITT) population, last observation carried forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | SNF472 300 mg | SNF 472 600 mg | SNF 472 Combined Dose Groups | Matching Placebo
Number analyzed (Participants) | 77 | 65 | 142 | 77
Participants | 46 | 41 | 87 | 37

5. Secondary Outcome: Number of Subjects With >=15% Progression in CAC Agatston Score at Week 52 for Each Dose Group and the Combined Dose Groups vs Placebo
Description: Agatston score is a semi-automated tool to calculate a score the reflects the extent of coronary artery calcification as detected by an unenhanced CT scan. Scores range from 0 to >1000 Agatston units where higher scores indicate an increased amount of calcification and an increased risk for a major adverse cardiac event. Change in Agatston Score values from baseline to Week 52 was calculated as a percentage of change (progression or worsening of calcification). The number of subjects with >=15% progression were counted for each treatment group, the combined treatments groups and placebo.
Time Frame: Baseline (Week 1, Day 1) and Week 52
Population: Modified intent-to-treat (mITT) population, last observation carried forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | SNF472 300 mg | SNF 472 600 mg | SNF 472 Combined Dose Groups | Matching Placebo
Number analyzed (Participants) | 77 | 65 | 142 | 77
Participants | 31 | 24 | 55 | 40

6. Secondary Outcome: Change in Log Thoracic Aorta Calcification Volume Score Between Baseline and Week 52 for Each Dose Group (300 mg and 600 mg) vs Placebo and the Combined Dose Groups vs Placebo
Description: Coronary Artery Calcification (CAC) Volume Score is a calculation to quantify the calcification of coronary artery calcium without factoring in the calcium density as measured by the CAC Agatston Score. The CAC volume score observed in the thoracic aorta was used for this analysis. The CAC volume Score was log-transformed and the primary outcome measure was the change in Log CAC Volume Score from Baseline to Week 52 for the combined dose groups and each dose group vs placebo. The secondary analysis used an ANCOVA model with the change in log volume score (log 52-week volume score - log baseline volume score) as the dependent variable and with a fixed effect term for the combined randomized treatment groups and log CAC volume score at baseline as a covariate. The least squares means for the treatment groups was estimated and back transformed.
  A smaller change from baseline to follow up is a better outcome.
Time Frame: Baseline (Week 1, Day 1) and Week 52
Population: Modified intent-to-treat (mITT) population, last observation carried forward (LOCF)
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | SNF472 300 mg | SNF 472 600 mg | SNF 472 Combined Dose Groups | Matching Placebo
Number analyzed (Participants) | 74 | 60 | 134 | 75
ratio | 1.25 [1.156 to 1.346] | 1.21 [1.113 to 1.318] | 1.23 [1.161 to 1.302] | 1.28 [1.187 to 1.381]

7. Secondary Outcome: Change in Log Thoracic Aorta Calcification Agatston Score Between Baseline and Week 52 for Each Dose Group (300 mg and 600 mg) vs Placebo and the Combined Dose Groups vs Placebo
Description: Coronary Artery Calcification (CAC) Agatston Score is a semi-automated tool to calculate a score that reflects the extent of coronary artery calcification as detected by an unenhanced CT scan. Scores range from 0 to >1000 Agatston units where higher scores indicate an increased amount of calcification and an increased risk for a major adverse cardiac event. This secondary outcome measure was the change in CAC Agatston Score in the thoracic aorta from Baseline to Week 52 for each dose group and the treated arms combined vs placebo. The analysis used an ANCOVA model with the change in log score (log 52-week score - log baseline score) as the dependent variable and with a fixed effect term for each randomized treatment groups and log CAC score at baseline as a covariate. The least squares means for each of the treatment groups separately and combined was estimated and back transformed. A smaller change from baseline to follow up is a better outcome.
Time Frame: Baseline (Week 1, Day 1) and Week 52
Population: Modified intent-to-treat (mITT) population, last observation carried forward (LOCF)
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | SNF472 300 mg | SNF 472 600 mg | SNF 472 Combined Dose Groups | Matching Placebo
Number analyzed (Participants) | 74 | 60 | 134 | 75
ratio | 1.30 [1.186 to 1.432] | 1.28 [1.149 to 1.416] | 1.29 [1.201 to 1.384] | 1.32 [1.205 to 1.452]

8. Secondary Outcome: Change in Log Aortic Valve Calcification Volume Score Between Baseline and Week 52 for Each Dose Group (300 mg and 600 mg) vs Placebo and the Combined Dose Groups vs Placebo
Description: Coronary Artery Calcification (CAC) Volume Score is a calculation to quantify the calcification of coronary artery calcium without factoring in the calcium density as measured by the CAC Agatston Score. The CAC volume score observed in the aortic valve was used for this analysis. The CAC volume Score was log-transformed and the primary outcome measure was the change in Log CAC Volume Score from Baseline to Week 52 for the combined dose groups and each dose group vs placebo. The secondary analysis used an ANCOVA model with the change in log volume score (log 52-week volume score - log baseline volume score) as the dependent variable and with a fixed effect term for the combined randomized treatment groups and log CAC volume score at baseline as a covariate. The least squares means for the treatment groups was estimated and back transformed.
  A smaller change from baseline to follow up is a better outcome.
Time Frame: Baseline (Week 1, Day 1) and Week 52
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | SNF472 300 mg | SNF 472 600 mg | SNF 472 Combined Dose Groups | Matching Placebo
Number analyzed (Participants) | 75 | 63 | 138 | 69
ratio | 1.28 [1.143 to 1.426] | 1.01 [0.899 to 1.144] | 1.14 [1.048 to 1.235] | 1.98 [1.768 to 2.226]

9. Secondary Outcome: Change in Log Aortic Valve Calcification Agatston Score Between Baseline and Week 52 for Each Dose Group (300 mg and 600 mg) vs Placebo and the Combined Dose Groups vs Placebo
Description: Coronary Artery Calcification (CAC) Agatston Score is a semi-automated tool to calculate a score the reflects the extent of coronary artery calcification as detected by an unenhanced CT scan. Scores range from 0 to >1000 Agatston units where higher scores indicate an increased amount of calcification and an increased risk for a major adverse cardiac event. This secondary outcome measure was the change in Log CAC Agatston Score or the aortic valve from Baseline to Week 52 for each dose group and the treated arms combined vs placebo. The analysis used an ANCOVA model with the change in log score (log 52-week score - log baseline score) as the dependent variable and with a fixed effect term for each randomized treatment groups and log CAC score at baseline as a covariate. The least squares means for each of the treatment groups separately and combined was estimated and back transformed. A smaller change from baseline to follow up is a better outcome.
Time Frame: Baseline (Week 1, Day 1) and Week 52
Population: Modified intent-to-treat (mITT) population, last observation carried forward (LOCF)
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | SNF472 300 mg | SNF 472 600 mg | SNF 472 Combined Dose Groups | Matching Placebo
Number analyzed (Participants) | 75 | 63 | 138 | 69
ratio | 1.33 [1.141 to 1.541] | 0.98 [0.836 to 1.160] | 1.14 [1.022 to 1.277] | 2.86 [2.449 to 3.349]

10. Secondary Outcome: Number of Participants With the Composite Safety Endpoint (Cardiovascular Death, Nonfatal Myocardial Infarction, Non-fatal Stroke, Heart Failure or Non-fatal Cardiac Arrest.
Description: The number of subjects meeting this composite safety endpoint were counted and expressed by the randomized arm as a % of patients for the safety population.terms resulting in death from cardiovascular causes, myocardial infarction, stroke, or heart failure for each dose group and placebo were summarized .
Time Frame: Baseline (Week 1, Day 1) and Week 52
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | SNF472 300 mg | SNF 472 600 mg | SNF 472 Combined Dose Groups | Matching Placebo
Number analyzed (Participants) | 92 | 91 | 183 | 90
Participants | 7 | 6 | 13 | 10

11. Secondary Outcome: Mortality Rate (All-cause) for Each Dose Group and Placebo
Description: The number of deaths were counted and expressed by the randomized arm as a % of patients for the safety population.
Time Frame: Baseline (Week 1, Day 1) and Week 52
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | SNF472 300 mg | SNF 472 600 mg | SNF 472 Combined Dose Groups | Matching Placebo
Number analyzed (Participants) | 92 | 91 | 183 | 90
Participants | 1 | 6 | 7 | 5

ADVERSE EVENTS:
Time Frame: Collected over one year
Arm/Group | SNF472 300 mg | SNF 472 600 mg | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 1/92 | 6/91 | 5/90
Serious Adverse Events (participants affected / at risk) | 38/92 | 55/91 | 49/90
Other Adverse Events (participants affected / at risk) | 62/92 | 64/91 | 67/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SNF472 300 mg (N=92) | SNF 472 600 mg (N=91) | Matching Placebo (N=90)
Pneumonia (Infections and infestations) | 4 (4) | 3 (3) | 7 (7)
Sepsis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Arteriovenous graft site infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Arteriovenous graft site abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Emphysematous cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vascular access site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection pseudomonas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Renal Transplant (Surgical and medical procedures) | 6 (6) | 14 (14) | 11 (11)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous graft aneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 3 (3) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 4 (4)
Cardiac arrest (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ulcerative gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Foreign body embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Calciphylaxis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Uraemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic ischaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cardiac stress test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Influenza a virus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Myocardial necrosis marker increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Stress echocardiogram abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lymphadenectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Toe amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SNF472 300 mg (N=92) | SNF 472 600 mg (N=91) | Matching Placebo (N=90)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 11 (11) | 10 (10)
Abdominal pain upper (Gastrointestinal disorders) | 11 (11) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 8 (8) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 5 (5) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7) | 7 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4) | 6 (6)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 9 (9) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT02966028/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT02966028/SAP_001.pdf